CLINICAL TRIAL: NCT00234650
Title: Evaluation of the Effect of Position Change During the Withdrawal Phase of Colonoscopy on Adenoma Detection Rate
Brief Title: Adenoma Detection Rate With Position Change at Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London North West Healthcare NHS Trust (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: 05/CO05/15
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Last update posted 2009-04-02 (Estimated); Status verified 2008-12

CONDITIONS: Polyps
Keywords: position change; adenoma; colonoscopy
MeSH Terms: conditions — Polyps; Adenoma | interventions — Colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy

SUMMARY:
The hypothesis to be tested is that position changes during the withdrawal phase of colonoscopy leads to a higher adenoma (polyp) detection rate because of better distension of the colon. Since adenomas are precancerous lesions the enhanced adenoma detection will increase the success of colorectal cancer screening programmes. This study will provide evidence for the value of position changes and encourage endoscopist to adopt position change as a routine in their practice.

May 2007: protocol amendment to include additional prospective analysis using High Definition TV (HDTV).

DETAILED DESCRIPTION:
Colorectal cancer is the second commonest cause of cancer death. In a majority of cases it is preceded by a precancerous lesion called an adenoma (commonly known as polyp). Detection and removal of adenomas at colonoscopy has been shown to reduce mortality from colorectal cancer. The success of the impending colorectal cancer screening programme to reduce cancer mortality in an average-risk population depends on optimal adenoma detection at colonoscopy. The detection of adenomas has been shown to vary between different endoscopist. Some of the factors that have been reported to affect adenoma detection rates included the time spent viewing, the adequacy of the bowel preparation and the time spent cleaning the colonic mucosa of excess fluid. Careful examination of proximal side of flexures, folds and valves by the endoscopist is equally important. However, even with careful examination adenoma detection rates have been shown to vary between endoscopist from 8.6% to 15.9%. Previous experience and training may be contributed to this difference. Some endoscopist adopt regular changes in position during the procedure to maximize distension of the colon. Better luminal distension enhances mucosal views for detection of the smaller adenomas. The validity of this approach has never been tested and we propose that this factor may contribute to the differences in adenoma detection rates.

Patients will be randomised to either position 1 first then position 2 or vice versa and examined twice. During one withdrawal the colon will be examined with the participant in the left lateral position only (position 1) or with position changes (position 2)or vice versa.

May 2007: protocol amendment to include additional prospective analysis using High Definition TV (HDTV). No further patient data collection involved.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred ot colonoscopy, age between 50 - 70 years

Exclusion Criteria:

* Patients with colorectal cancer, previous colonic surgery, active colitis and musculoskeletal problems Patients may also be excluded after the first insertion, if painful, routine care will proceed

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2005-10; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
adenoma detection rate for position 1 compared to position 2

SECONDARY OUTCOMES:
percentage of adenomas detected in all the participants for each position

CONTACTS AND LOCATIONS:
Overall Officials: Brian Saunders, MD, Principal Investigator — St Mark's Hospital, North West London NHS Trust
Locations (1):
- North West London NHS Trust, London, Middlesex, United Kingdom

REFERENCES:
- [Derived] East JE, Bassett P, Arebi N, Thomas-Gibson S, Guenther T, Saunders BP. Dynamic patient position changes during colonoscope withdrawal increase adenoma detection: a randomized, crossover trial. Gastrointest Endosc. 2011 Mar;73(3):456-63. doi: 10.1016/j.gie.2010.07.046. Epub 2010 Oct 15. PMID 20950801